CLINICAL TRIAL: NCT02010450
Title: Re-enforcing Safe Sleep Practices for Caregivers With Tangible Incentives: Pilot Testing of the MSSC Physician Safe Sleep Taskforce Caregiver Incentive Toolkit
Brief Title: Re-enforcing Safe Sleep Practices for Caregivers With Tangible Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-017
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Safe Sleep Education
Keywords: Sudden Infant Death Syndrome; SIDS; safe sleep; safe sleep message
MeSH Terms: conditions — Sudden Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wearable Blanket (Experimental): subjects randomized to this group will receive a wearable blanket (sleep sack) that contains a safe sleep message.
  Interventions: Other: Wearable Blanket (Sleep Sack)
- Control Group (Active Comparator): subjects randomized to this group will receive an incentive item (such as a University of Kansas Pediatrics water Bottle) that does not contain the safe sleep message.
  Interventions: Other: Incentive Item

INTERVENTIONS:
Other: Wearable Blanket (Sleep Sack)
  Arms: Wearable Blanket
Other: Incentive Item
  Arms: Control Group

SUMMARY:
This study is a pilot study to test the effectiveness of incentive items to increase compliance of infant safe sleep practices among caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Parent of 1-month old baby
* Over the age of 18
* Be able to speak and read English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
dichotomous sleep variable (safe vs unsafe) | Change from Baseline to 2 Months
  change measured using "safe sleep quiz" questionnaire

SECONDARY OUTCOMES:
determine which incentive item provided is most effective in reinforcing the safe sleep message | Change from Baseline to 2 Months
  determination to be assessed using questionnaire completed by caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn R Ahlers-Schmidt, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- KU Wichita Pediatrics, Wichita, Kansas, United States